CLINICAL TRIAL: NCT03003585
Title: Comparison of Effects of Direct Laryngoscopic and Fiberoptic Oral Endotracheal Intubation on Intraocular Pressure
Brief Title: Effects of Direct Laryngoscopic and Fiberoptic Intubation on Intraocular Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ahmet Selim Ozkan, M.D., Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Asozkan-2
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Intraocular Pressure; Intubation Complication
Keywords: intraocular pressure; direct laryngoscopy; fiberoptic bronchoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fiberoptic bronchoscopy (Active Comparator): Evaluate the difference between the two groups about hemodynamic and intraocular pressure responses.
  Interventions: Other: Fiberoptic bronchoscope
- Direct laryngoscopy (Active Comparator): Evaluate the difference between the two groups about hemodynamic and intraocular pressure responses.
  Interventions: Other: Direct laryngoscope

INTERVENTIONS:
Other: Direct laryngoscope — This device is used in endotracheal intubation and tonopen device for measuring of intraocular pressure. The investigators want to evaluate which one is better.
  Arms: Direct laryngoscopy
Other: Fiberoptic bronchoscope — This device is used in endotracheal intubation and tonopen device for measuring of intraocular pressure. The investigators want to evaluate which one is better.
  Arms: Fiberoptic bronchoscopy

SUMMARY:
In this study, the investigators aimed to compare the effects of direct laryngoscopic and fiberoptic endotracheal intubation on intraocular pressure.

DETAILED DESCRIPTION:
Material and Method: Total of 54 American Society of Anesthesiologist Grade 1-2, Mallampati score 1 or 2, age between 18 to 65 patient planned to undergo nonopthalmic surgery will be included to study. Patients with glaucoma, diabetes mellitus, cardiovascular and pulmonary diseases, American Society of Anesthesiologist Grade III and IV, body mass index more than 35, difficult intubation, undergo obstetrical surgery and propofol, fentanyl, rocuronium contraindicated will be excluded from the study. Patients will be divided randomly into 2 groups as direct laryngoscopic and fiberoptic intubation group. Patients will be preoxygenated with %100 O2 for 3 minutes then anesthesia will be induced using propofol 2 mg / kg, fentanyl 1 mcg/kg, and rocuronium 0,5 mg / kg in both groups. After 3 minutes mask ventilation, patients will be intubated (women with No:7-7,5, men with No:8-8,5 intubation tube). Systolic blood pressure, diastolic blood pressure, mean arterial pressure, peripheral oxygen saturation,perfusion index will be recorded and intraocular pressure measured by ophthalmologist by tonopen device will be recorded pre-induction (basal), after induction, 1,2,3,5 minutes after intubation, respectively. Period between handling of laryngoscope or fiberoptic device after termination of mask ventilation and obtain end tidal CO2 will be accepted as application time and recorded. Study will be terminated after 5th minute values taken.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologist) Grade 1-2,
* Mallampati score 1 or 2,
* Age between 18 to 65
* Patient planned to undergo nonopthalmic surgery.

Exclusion Criteria:

* Patients with glaucoma, diabetes mellitus, cardiovascular and pulmonary diseases, ASA Grade III and IV, BMI more than 35,
* Patients with difficult intubation,
* Patients undergoing obstetrical surgery and propofol, fentanyl, rocuronium contraindicated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-12; Primary Completion 2017-02 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | From Beginning of Anesthesia induction to 5th minutes of intubation
Heart rate | From Beginning of Anesthesia induction to 5th minutes of intubation
Adverse events | within the first 24 hour after surgery
Intraocular pressure | From Beginning of Anesthesia induction to 5th minutes of intubation